CLINICAL TRIAL: NCT02968199
Title: Development of a Community-based Network to Promote Smoking Cessation Among Female Smokers in Hong Kong
Brief Title: Building a Community-based Network to Promote Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Smoking_1
Record Dates: First submitted 2016-11-16; First posted 2016-11-18 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Smoking
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Masking Description: The study was not a randomized controlled trial. Participants and outcome assessors were not blinded.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Referred women (Experimental): A brief intervention based on the'5 A' model developed by the Agency for Health Care Policy and Research in the United States.
  Interventions: Behavioral: A brief intervention

INTERVENTIONS:
Behavioral: A brief intervention — The content of the intervention includes: (1) asking about tobacco use; (2) advising cessation; (3) assessing willingness to quit; (4) assisting in the attempt to quit; and (5) arranging follow-up.

SUMMARY:
This study describes the development of a community-based network to promote smoking cessation among female smokers in Hong Kong.

DETAILED DESCRIPTION:
There is growing concern about the use of tobacco among women in Hong Kong. Nevertheless, nearly all of them reported that they had not attended smoking cessation services provided by the government and other organizations, of which only 6.7% indicated that they would like to attend, demonstrating the need for population-based smoking cessation interventions targeting female smokers in Hong Kong. In response to the increased number of female smokers and their low usage rates of smoking cessation services, the first smoking cessation hotline for female smokers in Hong Kong was established in 2006 by the University of Hong Kong. The aim of this study was to describe the development of a community-based network to promote the smoking cessation hotline among female smokers in Hong Kong.

ELIGIBILITY:
Inclusion Criteria:

* Female Hong Kong Chinese current smokers
* Aged 15 years or above
* Able to speak and understand Cantonese
* Willing to receive face-to-face or telephone counseling

Exclusion Criteria:

* Those who were participating in other smoking cessation programs or services

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 457 (Actual)
Dates: Start 2006-01 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
self-reported 7-day point prevalence of abstinence | 6 months

SECONDARY OUTCOMES:
self-reported reduction of ≥ 50% in cigarette consumption | 6 months
Levels of self-efficacy at baseline | baseline
Levels of self-efficacy at six months | six months

CONTACTS AND LOCATIONS:
Overall Officials: William, Ho Cheung LI, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong SAR, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li WH, Chan SS, Wan ZS, Wang MP, Ho KY, Lam TH. Development of a community-based network to promote smoking cessation among female smokers in Hong Kong. BMC Public Health. 2017 Apr 11;17(1):311. doi: 10.1186/s12889-017-4213-z. PMID 28399845